CLINICAL TRIAL: NCT05304208
Title: Phase I, Open-Label Study With Dendritic Cell Therapy (MesoPher) In Combination With Ex-tended-Pleurectomy/Decortication After Chemotherapy in Subjects With Resectable Mesothelioma
Brief Title: dENdritic Cell Therapy Combined With SURgEry in Mesothelioma
Acronym: ENSURE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Joachim Aerts, MD PhD, Professor, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 76712
Record Dates: First submitted 2022-01-20; First posted 2022-03-31 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Mesotheliomas Pleural
Keywords: dendritic cell therapy; malignant pleural mesothelioma; mesopher; pleurectomy/decortication
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Before standard-of-care chemotherapy, a leukapheresis will be performed and monocytes will be used for differentiation to DCs using specific cytokines. Allogeneic tumor lysate (Pheralys) loaded autologous DCs (MesoPher) will be re-injected 3 weeks after completing chemotherapy, 2 times every other week. Four weeks after the first injection with DCT, patients will undergo eP/D surgery and receive three bi-weekly injections with DCT (starting 4 weeks after surgery). If there is a surplus of vaccinations, a 6th and 7th vaccination at 3 and six months after the last vaccination could be considered by the treating physician.
  Interventions: Biological: Mesopher

INTERVENTIONS:
Biological: Mesopher — autologous monocyte-derived DCs loaded with PheraLys (tumor cell lysate)

SUMMARY:
The ENSURE trial is an open label, single center, phase 1, feasibility study. Sixteen adult patients diagnosed with resectable epithelioid malignant pleural mesothelioma (MPM) will be enrolled following first-line chemotherapy. Before standard-of-care chemotherapy, a leukapheresis will be performed and monocytes will be used for differentiation to dendritic cells (DCs) using specific cytokines. Allogeneic tumor lysate (Pheralys) loaded autologous DCs (MesoPher) will be re-injected 3 weeks after completing chemotherapy, 2 times every other week. Four weeks after the first injection with dendritic cell therapy (DCT), patients will undergo extrapleural pleurectomy/decortication (eP/D) surgery and receive three bi-weekly injections with DCT (starting 4 weeks after surgery). In total, five DC vaccinations will be administered. A tumor biopsy will be collected before starting neo-adjuvant DCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of epithelioid MPM who are eligible for 2 to 4 cycles of platinum-based chemotherapy. Patients who progressed after chemotherapy will not be discontinued from the trial if they are still eligible for eP/D and none of the exclusion criteria is present (e.g. local progression with only focal chest invasion).
* Patients must be at least 18 years old and must be able to give written informed con-sent.
* Resectable disease defined by stage cT1-3, N0-1, M0 (I to IIIA) according to UICC TNM classification (8th edition). A fluorodeoxyglucose (FDG)-positron emission tomography (PET)-computerized tomography (CT) scan with fusion images showing absence of M1, N2 involvement is required. Focal chest wall lesions are acceptable.
* Tumor tissue available after completing chemotherapy and before starting treatment with DCT. Tumor tissue can be obtained by either a CT-guided needle biopsy or a Video-assisted thoracoscopic surgery (VATS) biopsy.
* Fit to receive platinum-based chemotherapy (as per standard of care of the treating physician/Institution) and undergo a P/D with optional removal of hemidiaphragm and pericardium. The responsible surgeon and chest physician should judge the required fitness prior to registration, taking into account the results of all the relevant (i.e. pulmonary, cardiac) examinations.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Appendix 2).
* Ability to return to the study center for adequate follow-up and vaccinations.
* Positive delayed-type hypersensitivity (DTH) skin test (induration > 2mm after 48 hrs) against at least one positive control antigen tetanus toxoid.
* Written informed consent according to ICH-GCP.
* Subjects must have adequate organ function and adequate bone marrow reserve at screening:

  * creatinine ≤ 1.5 × upper limit of normal [ULN] or glomerular filtration rate ≥ 50 mL/min
  * alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin ≤ 1.5 × ULN
  * Absolute neutrophil count ≥1.5 x 109/L, platelet count ≥100 x 109/L, and Hb ≥9.0 g/dL. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test just prior to the first study drug administration on Day 1, and must be willing to use an effective contraceptive method (intrauterine devices, hormonal contraceptives, contraceptive pill, implants, transdermal patches, hormonal vaginal devices, infusions with prolonged release) or true abstinence (when this is in line with the preferred and usual lifestyle)* during the study and for at least 12 months after the last study drug administration.

  *True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (such as calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Men must be willing to use an effective contraceptive method (e.g. condom, vasectomy) during the study and for at least 12 months after the last study drug administration.
* Written informed consent according to the International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP) guidelines.

Exclusion Criteria:

* Clinical or radiological invasion of mediastinal structures (heart, aorta, spine, esophagus, etc.) and widespread chest wall invasion (stage T4). Involvement of N2 nodes. Stage IV (metastatic disease).
* Any different histology from the epithelioid MPM (as per assessed at time of diagnosis).
* Unavailability of tumor tissue after completing chemotherapy and before starting treatment with DCT.
* Subject with any concurrent medical, psychological or psychiatric disease or condition that is likely to compromise the ability to give informed consent or to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
* Use of >10 mg of prednisolone or equivalent/day (or other immunosuppressive agents) during the past 6 weeks before the first study drug administration and throughout the study. Prophylactic usage of dexamethasone (steroids) during chemotherapy is excluded from this 6-week interval. Inhaled or topical steroids, and adrenal replacement steroid ≤10 mg daily prednisone equivalent, are permit-ted in the absence of active autoimmune disease.
* Major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery (other than eP/D) during the course of study treatment.
* Subject with any previous malignancy except adequately treated basal cell or squamous cell skin cancer, superficial or in-situ cancer of the bladder or other cancer for which the subject has been disease-free for at least 3 years.
* Prior treatment of any kind for mesothelioma, especially prophylactic track irradiation after diagnostic procedures.
* Clinically significant pleural effusion that cannot be managed with thoracentesis or pleurodesis (according to institutional practice). If pleurodesis is considered, it should be done before randomization.
* Subject with any known active serious infection, including human immunodeficiency virus (HIV), hepatitis B or C virus, or syphilis infection.
* Subject with a history of autoimmune disease, except for diabetes mellitus type I or other conditions, where patient can be eligible following discussion with medical monitor.
* Subject who has received an organ allograft.
* Serious intercurrent chronic or acute illness such as pulmonary (COPD or asthma) or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the study coordinator to constitute an unwarranted high risk for eP/D or investigational DCT.
* Pregnant women, nursing mothers, lactating women, and women of child-bearing potential who are unwilling to use effective contraceptive methods (intrauterine de-vices, hormonal contraceptives, contraceptive pill, implants, transdermal patches, hormonal vaginal devices, infusions with prolonged release) during the study and for at least 12 months after the last study drug administration.
* Men unwilling to use effective contraception for the duration of the study and for at least 12 months after the last study drug administration.
* Inadequate peripheral vein access to perform leukapheresis
* History of receiving any investigational treatment within 28 days of randomization.
* Absence of assurance of compliance with the protocol. Lack of availability for fol-low-up assessment.
* Patients with a known allergy to shellfish (may contain KLH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participant who are alive and have completed (neo)adjuvant DCT (5 administrations) and surgery at week 15 (+4 weeks) without extended treatment-related delay, persisting grade 3-4 treatment side-effects or evidence of progression [Feasibility] | 2 years
  To determine the feasibility of DCT with Mesopher performed before and after eP/D in patients with resectable epithelioid MPM who received first line chemotherapy. Feasibility is measured by the number of patient who are alive and have completed neo-adjuvant plus adjuvant DCT (5 administrations in total or less in case of production shortage) and surgery at week 15 (+4 weeks) without extended treatment-related delay, persisting grade 3- 4 treatment side-effects or evidence of progression/relapse. Patients who markedly progressed after chemotherapy will be discontinued from the trial and will be considered as failures for assessment of the primary end-point.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 [Safety and Tolerability] | 2 years
  To assess the safety of DCT with Mesopher performed before and after eP/D in patients with resectable epithelioid MPM.
Median progression free and median overall survival since start of treatment [Efficacy] | 2 years
  To evaluate the efficacy of combining DCT and eP/D after chemotherapy in patients with resectable epithelioid MPM. Efficacy is measured by median progression free and median overall survival since start of treatment.

OTHER OUTCOMES:
Number of participants with increased immune cell infiltration in tumor tissue induced by (neo)adjuvant DCT [Anti-tumor immune response] | 2 years
  To determine the anti-tumor immune response induced by (neo)adjuvant DCT. In order to analyze if DC-therapy induced a (tumor-specific) immune response, the following analyses will be performed:
  1. Evaluate immune cell infiltration in tumor tissue prior and post DCT.
  2. Characterize T-cell receptor (TCR) repertoire analysis of tumor-infiltrating T cells.
  3. Characterize tumor-specific and lysate specific IFNy production by IFNy ELISPOT assay.
  4. Characterize the phenotype of immune cell populations in the tumor and peripheral blood prior and post DCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided